CLINICAL TRIAL: NCT02077907
Title: Comparison of Four Different Supplementary Foods in the Treatment of Moderate Acute Malnutrition (MAM) in Children in Sierra Leone: a Cluster-randomised, Controlled Clinical Effectiveness Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Ebola virus disease outbreak
Sponsor: Tufts University (Other)
Collaborators: Washington University School of Medicine (Other); Project Peanut Butter (Other); United Nations World Food Programme (WFP) (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AID-016-Sierra Leone; USAID (Other Grant/Funding Number: AFP-C-00-09-00016-00)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Moderate Acute Malnutrition (MAM)
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Super Cereal Plus (SC+) (Active Comparator): 800 kcal/d, 215 g/d
  Current protocol for treating MAM is supplemental food distribution, often providing a fortified blended food (FBF) that requires cooking. In Sierra Leone, their FBF standard is Super Cereal Plus.
  Interventions: Dietary Supplement: Super Cereal Plus (SC+)
- Super Cereal (SC) and oil and sugar (Experimental): 200 g SC and 20 g fortified oil and 15 g sugar, per day
  Fortified blended food (FBF) Fortified Oil with Vitamins A & D
  Interventions: Dietary Supplement: Super Cereal (SC), fortified oil, sugar
- Corn Soy Blend 14 (CSB14) and fortified oil (Experimental): 978 kcal/day - 150 g CSB14 and 45 g oil, per day
  Fortified blended food (FBF) Fortified Oil with Vitamins A & D
  Interventions: Dietary Supplement: Corn Soy Blend 14 (CSB14) and fortified oil
- Plumpy'Sup (Experimental): 500 kcal/d, 92 g/d
  Ready-to-Use Supplementary Food (RUSF)
  Interventions: Dietary Supplement: Plumpy Sup

INTERVENTIONS:
Dietary Supplement: Super Cereal Plus (SC+)
  Arms: Super Cereal Plus (SC+)
Dietary Supplement: Super Cereal (SC), fortified oil, sugar
  Arms: Super Cereal (SC) and oil and sugar
Dietary Supplement: Plumpy Sup
  Arms: Plumpy'Sup
Dietary Supplement: Corn Soy Blend 14 (CSB14) and fortified oil
  Arms: Corn Soy Blend 14 (CSB14) and fortified oil

SUMMARY:
The objective of this study is to test and compare the effectiveness and cost-effectiveness of four supplementary foods for the treatment of moderate acute malnutrition (MAM) in normal programmatic settings in Sierra Leone. Study participants will receive one of four test foods varying in energy and nutrient density as well as amounts provided.

1. Super Cereal Plus (SC+) at 800 kcal/d, 215 g/d (Control group)
2. Super Cereal (SC) and oil and sugar at 998 kcal/d - 200 g SC and 20 g oil and 20 g sugar, per day
3. Corn-soy Blend 14 (CSB14) and oil at 978 kcal/day - 150 g CSB14 and 45 g oil, per day
4. Plumpy'Sup - 500 kcal/d, 92 g/d

This will be a prospective, randomised, controlled effectiveness trial.

Aims

1. (Impact) To compare the effectiveness of four supplementary foods in the treatment of moderate acute malnutrition (MAM) in normal programmatic settings in Sierra Leone.
2. (Cost) To estimate the relative cost-effectiveness (marginal cost per child recovered from MAM, relative to comparison group, SC+) of implementing the feeding program using each commodity, taking into consideration costs of procurement/production and distribution
3. (Process) To evaluate the determinants of effectiveness including: consumption adherence, preparation compliance, targeting/sharing of supplement, food components and preparation, adverse effects of foods, water contamination, hygiene and health behaviors, SES, food security, perceived barriers

Outcomes

1. Recovery from MAM

   1. Percent of children recovered from MAM (defined as achieving mid-upper arm circumference (MUAC) ≥ 12.5 cm by 12 weeks once)
   2. Percent default/non-response: children who do not recover after 12 weeks
   3. Percent relapse: children who become MAM again within 6 months of recovery
2. Mean number of weeks to recovery

Hypothesis The children with MAM fed Super Cereal and oil and sugar, CSB14 and oil or Plumpy'Sup will have similar recovery outcomes to those children fed Super Cereal Plus.

Null: The children with MAM fed Super Cereal and oil and sugar, CSB14 and oil or Plumpy'Sup will have different recovery outcomes to those children fed Super Cereal Plus.

ELIGIBILITY:
Beneficiary Children (Children 6 months to 59 months old)

Inclusion Criteria

* Child diagnosed with MAM and enrolled to receive a ration from a feeding site (i.e. enrolled in the SFP) Exclusion Criteria
* Children with bipedal oedema
* Children receiving food rations from another organization (e.g. USAID or UNICEF)

Beneficiary Mothers/Caretakers (Mothers/Caretakers of Children 6 months to 59 months old)

Inclusion Criteria

* Beneficiary Mother/Caretaker whose child is diagnosed with MAM and enrolled to receive a ration from a feeding site
* Beneficiary Mother/Caretaker has no age restrictions for inclusion (Note: Mothers/caretakers will be asked to participate regardless of age and consented appropriately; it is possible some mothers may be minors)
* Subject who is voluntarily willing to participate and indicates by signing (or marking with a thumbprint) the consent form.

Exclusion Criteria

• Beneficiary Mothers/Caretakers who participate in an interview, observation or FGD once for this study will not be eligible again for participation

Community Health Volunteers (CHV)/Health Development Committee Members (HDC) Inclusion Criteria

* Community Health Volunteers & Health Development Committee Members serving within the catchment area for the PHUs
* Community Health Volunteers that have been present during the study period
* Subject who is voluntarily willing to participate and indicates by signing the consent form

PPB and Clinic Staff Members Inclusion Criteria

* All staff members from Project Peanut Butter and the PHU who are directly involved in the feeding program
* Subject who is voluntarily willing to participate and indicates by signing the consent form Exclusion Criteria
* Staff members who joined too recently to have experience of the program change (new commodities)

Village Elders/Headmen Inclusion Criteria

* Village elder/headmen in study commune
* Subject who is voluntarily willing to participate and indicates by signing the consent form Exclusion Criteria
* Village elder/headmen whose community is not involved in the feeding program

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1147 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Recovery from MAM | 12 weeks
  1. Percent of children recovered from MAM (defined as achieving mid-upper arm circumference (MUAC) ≥ 12.5 cm by 12 weeks once)
  2. Percent default/non-response: children who do not recover after 12 weeks
  3. Percent relapse: children who become MAM again within 6 months of recovery

SECONDARY OUTCOMES:
Change in Growth rates | 12 weeks
  Subjects will return to clinic every 2 weeks until MUAC of 12.5 cm is reached or until 12 weeks has elapsed. Follow-up recovery will then be measured at 6 months. At each clinic visit growth will be measured.
Duration of treatment | 12 weeks
  Subjects will return to clinic every 2 weeks until MUAC of 12.5 cm is reached or until 12 weeks has elapsed. Follow-up recovery will then be measured at 6 months. Time to achieve MUAC of 12.5 cm will be documented.
Cost estimates for participation | 12 weeks
  Average cost of treatment will be measured per participant, this includes intervention costs and any medical costs needed by participants. The study costs no money to participants.
Default reason | 12 weeks
  If a child defaults, then the reason will be an outcome measure. Reasons to default include loss to follow-up (the child will be attempted to be contacted 3 times prior to being considered lost), death, or he/she enters into the inpatient clinic.
Change in recovery status after 12 weeks | 6 months
  Any changes in recovery will be measured at 6 months at follow-up visits

OTHER OUTCOMES:
Relative cost-effectiveness | 12 weeks
  To estimate the relative cost-effectiveness (marginal cost per child recovered from MAM, relative to comparison group, SC+) of implementing the feeding program using each commodity, taking into consideration costs of procurement/production and distribution
Determinants of effectiveness | 12 weeks
  To evaluate the determinants of effectiveness including: consumption adherence, preparation compliance, targeting/sharing of supplement, food components and preparation, adverse effects of foods, hygiene and health behaviors, SES, food security, perceived barriers

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine; Beatrice Rogers, PhD, Principal Investigator — Tufts University, Friedman School of Nutrition